CLINICAL TRIAL: NCT01213979
Title: Open-label Pharmacokinetic Study of Iron Isomaltoside 1000 (Monofer®) Administered by 500 mg IV Bolus Injection or 1000 mg Intravenous Infusion to Patients With Non-hematological Malignancies Associated With Chemotherapy Induced Anaemia (CIA)(PK-CIA-04)
Brief Title: Open-label Pharmacokinetic Study of Iron Isomaltoside 1000 (Monofer®) Administered by 500 mg IV Bolus Injection or 1000 mg Intravenous Infusion to Patients With Non-hematological Malignancies Associated With Chemotherapy Induced Anaemia (CIA)
Acronym: PK-CIA-04
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmacosmos A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-Monofer-PK-CIA-04
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Non-hematological Malignancies
MeSH Terms: interventions — iron isomaltoside 1000

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1000 mg iron isomaltoside 1000 as intravenous infusion (Active Comparator)
  Interventions: Drug: 1000 mg iron isomaltoside 1000
- 500 mg iron isomaltoside 1000 as bolus injection (Active Comparator)
  Interventions: Drug: 500 mg iron isomaltoside 1000

INTERVENTIONS:
Drug: 500 mg iron isomaltoside 1000 — 500 mg iron isomaltoside 1000 given as a bolus injection over 2 minutes
  Arms: 500 mg iron isomaltoside 1000 as bolus injection
Drug: 1000 mg iron isomaltoside 1000 — 1000 mg iron isomaltoside 1000 given as a infusion over 15 minutes
  Arms: 1000 mg iron isomaltoside 1000 as intravenous infusion

SUMMARY:
The purpose of this study is to assess the pharmakokinetic properties of higher doses (500 mg and 1000 mg) of Monofer(R)in patients suffering from non-hematological malignancies with Chemotherapy induced anaemia.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged more than 18 years.
2. Weight above 50 kg.
3. Subjects diagnosed with non-hematological malignancies (solid tumors only) receiving chemotherapy at least 1 day prior to screening and who are going to receive at least two more chemotherapy cycles.
4. Hb < 12 g/dL.
5. TfS <50%.
6. Serum Ferritin <800 ng/ml.
7. An Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
8. Willingness to participate after informed consent.

Exclusion Criteria:

1. Anaemia caused primarily by other factors than CIA.
2. IV or oral iron treatment within 4 weeks prior to screening visit.
3. Erythrypoietin treatment within 4 weeks prior to screening visit.
4. Blood transfusion within 4 weeks prior to screening visit.
5. Imminent expectation of blood transfusion on part of treating physician.
6. Iron overload or disturbances in utilization of iron (e.g. haemochromatosis and haemosiderosis).
7. Drug hypersensitivity (i.e. previous hypersensitivity to Iron Dextran or iron mono- or disaccharide complexes or to iron sulfate).
8. Known hypersensitivity to any excipients in the investigational drug products.
9. Subjects with a history of multiple allergies.
10. Decompensated liver cirrhosis and hepatitis (alanine aminotransferase (ALAT) > 3 times upper normal limit).
11. History of Immunocompromise and/or history of Hepatitis B and/or C.
12. Active acute or chronic infections (assessed by clinical judgement and if deemed necessary by investigator supplied with white blood cells (WBC) and C-reactive protein (CRP)).
13. Rheumatoid arthritis with symptoms or signs of active joint inflammation.
14. Pregnancy and nursing (To avoid pregnancy, women have to be postmenopausal (at least 12 months must have elapsed since last menstruation), surgically sterile, or women of child bearing potential must use one of the following contraceptives during the whole study period and after the study has ended for at least 5 times plasma biological half-life (5 days) of the investigational medicinal product: Contraceptive pills, intrauterine devices (IUD), contraceptive depot injections (prolonged-release gestagen), subdermal implantation, vaginal ring, and transdermal patches).
15. Planned elective surgery during the study.
16. Participation in any other clinical study (except chemotherapy protocol) within 3 months prior to screening.
17. Known intolerance to oral iron treatment.
18. Untreated B12 or folate deficiency.
19. Any other medical condition that, in the opinion of Principal Investigator, may cause the subject to be unsuitable for the completion of the study or place the subject at potential risk from being in the study. Example, Uncontrolled Hypertension, Unstable Ischemic Heart Disease or Uncontrolled Diabetes Mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-02; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Total serum iron pharmakokinetic parameters | 24, 48 and 72 hours